CLINICAL TRIAL: NCT02532374
Title: A Single-center, Open-label, Ascending Nicotine Levels Study to Investigate the Nicotine Pharmacokinetic and Pharmacodynamics Profiles, Safety and Tolerability of P3L in Smoking Healthy Subjects in Relation to Nicorette® Inhalator
Brief Title: Nicotine Pharmacokinetic and Pharmacodynamics Profile, Safety and Tolerability of P3L
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philip Morris Products S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: P3L-PK-01-NZ; P3L-PK-01-NZ (Other: Philip Morris Products S.A)
Record Dates: First submitted 2015-08-21; First posted 2015-08-25 (Estimated); Results first posted 2017-06-15 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Smoking
Keywords: nicotine absorption; nicotine containing product; adult smoker; Nicorette; nicotine delivery system
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nicorette® inhalator then P3L (Experimental): Each subject will use the Nicorette® inhalator (15 mg) on Visit 3, and then use the P3L aerosol at nicotine dose levels of approximately 50 µg/puff, 80 µg/puff and 150 µg/puff on Visits 4, 5 and 6, respectively.
  Interventions: Other: Nicorette® inhalator; Other: P3L

INTERVENTIONS:
Other: Nicorette® inhalator — Subjects will inhale the Nicorette® inhalator (15 mg) at the rate of one deep inhalation every 15 seconds on average, over approximately 20 minutes (80 inhalations in total).
Other: P3L — Subjects will inhale P3L (50 µg/puff, 80 µg/puff and 150 µg/puff) at the rate of one inhalation every 30 seconds on average, over approximately 6 minutes (i.e., 12 inhalations in total).

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics (PK) and pharmacodynamics (PD, i.e., subjective effects) profiles, and the safety and tolerability of the nicotine-containing aerosol delivered by Platform 3 Liquid (P3L) system at three different nicotine levels in smoking healthy subjects in relation to Nicorette® inhalator.

DETAILED DESCRIPTION:
The entire study will last between 16 to 49 days per subject. This includes :

* a screening period of up to 4 weeks prior to admission,
* 1 day of admission (Visit 2): after all inclusion/exclusion criteria are checked, all eligible subjects will be enrolled and perform a product test, first with P3L (at nicotine dose levels of approximately 50 μg/puff) and subsequently with Nicorette® inhalator (3 to 5 inhalations for each product).
* 4 days of on-site product use (one day with Nicorette® inhalator [Visit 3] and three days with P3L [Visit 4, Visit 5 and Visit 6]),
* 1 to 3 days between each product use and
* a 7-day safety follow-up period (discharge + 7 days), during which there are no scheduled investigational visits, and during which adverse events (AEs) and serious adverse events (SAEs) can be spontaneously reported by the subjects and the follow-up of AEs/SAEs will be conducted by the study investigational site.

Subjects will come to the investigational site the night before each assessment day, at least 12 hours prior to the product use, on Visit 4, Visit 5, and Visit 6. Subjects will stay overnight at the investigational site between the admission visit (Visit 2) and Visit 3. Smoking or use of any tobacco/nicotine-containing products or electronic cigarettes, apart from product use assigned on the assessment days, will not be allowed during their stay at the investigational site. Smoking will be allowed once the subjects have left the investigational site.

The maximum concentration of nicotine (Cmax) and the area under the concentration-time curve from start of product use to the last quantifiable time point (AUC0-last) will be derived from multiple blood sampling pre- and post-product use, and corrected for baseline nicotine concentration.

ELIGIBILITY:
Inclusion Criteria:

* Subject is Caucasian
* Smoking, healthy subject as judged by the Investigator
* Subject smoked at least 10 commercially available non-menthol cigarettes (CCs) per day for the last 4 weeks
* Subject has smoked for at least the last 3 years prior to screening
* Subject does not plan to quit smoking in the next 3 months

Exclusion Criteria:

* As per Investigator judgment, the subject cannot participate in the study for any reason (e.g., medical, psychiatric, and/or social reason)
* Subject has donated or been in receipt of whole blood or blood products within 3 months prior to Admission Visit
* Female subject is pregnant or breast feeding
* Female subject does not agree to use an acceptable method of effective contraception
* Female subject uses estrogen-containing hormonal contraception or hormone replacement therapy

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-10; Primary Completion 2015-10 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christelle Haziza, PhD, Study Chair — Philip Morris Products S.A.; Chris Wynne, MD, Principal Investigator — Christchurch Clinical Studies Trust Ltd (CCST)
Locations (1):
- Christchurch Clinical Studies Trust Ltd (CCST), Christchurch, New Zealand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Teichert A, Brossard P, Felber Medlin L, Sandalic L, Franzon M, Wynne C, Laugesen M, Ludicke F. Evaluation of Nicotine Pharmacokinetics and Subjective Effects following Use of a Novel Nicotine Delivery System. Nicotine Tob Res. 2018 Mar 6;20(4):458-465. doi: 10.1093/ntr/ntx093. PMID 28482017

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study initiated (1st subject screened): 07 October 2015
  At admission, all the subjects were to try the P3L (50 μg/puff) and Nicorette® inhalator.
  Smoking or use of any tobacco/nicotine-containing products or electronic cigarettes, apart from product use assigned on the assessment days, was not allowed during the visits on site.
Pre-assignment Details: Enrolled population = 16 subjects
  All enrolled subjects met all of the inclusion and none of the exclusion criteria for the study.
Period: Overall Study
Arm/Group | Nicorette® Inhalator Then P3L
Started | 16
Nicorette Inhalator (Visit 3) | 15
P3L 50 μg/Puff (Visit 4) | 15
P3L 80 μg/Puff (Visit 5) | 14
P3L150 μg/Puff (Visit 6) | 14
Completed | 14
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: PK population: all the subjects who have signed the informed consent, completed at least one P3L product use period and for whom at least one PK parameter can been derived. No subjects were excluded due to major protocol deviations impacting the evaluation of the results.
  1 subject withdrew after the product test at the admission visit.
Arm/Group | Nicorette® Inhalator Then P3L
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.8 (13.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 8
Daily CC consumption at Screening [Count of Participants; unit: Participants]
  10 to 19 cig/day | 9
  > 19 cig/day | 6

OUTCOME MEASURES:

1. Primary Outcome: Maximum Concentration (Cmax) of Nicotine Following Single Use of Nicorette® Inhalator
Description: T0 = start of product use.
  Derived from multiple blood sampling pre- and post-product use on Visit 3 (over 240 minutes post-product use).
  Geometric Least Squares (geometric LS) means are provided.
Time Frame: Visit 3: blood taken at 45, 30 and 15 minutes prior to T0 and 2, 4, 7, 10, 15, 20, 30, 40, 50, 60, 120, and 240 minutes after T0.
Population: PK population: all the subjects who have signed the informed consent, completed at least one P3L product use period and for whom at least one PK parameter can been derived.
  => 16 subjects - 1 subject withdrew after the product test at the admission visit =15 subjects
Measure: Least Squares Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Nicorette® Inhalator
Number analyzed (Participants) | 15
ng/mL | 6.095 [4.243 to 8.755]

2. Primary Outcome: Maximum Concentration (Cmax) of Nicotine Following Single Use of P3L 50 µg/Puff
Description: T0 = start of product use.
  Derived from multiple blood sampling pre- and post-product use on Visit 4 (over 240 minutes post-product use).
  Geometric Least Squares (geometric LS) means are provided.
Time Frame: Visit 4: blood taken at 45, 30 and 15 minutes prior to T0 and 2, 4, 7, 10, 15, 20, 30, 40, 50, 60, 120, and 240 minutes after T0.
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: ng/mL
Groups:
- P3L 50 µg/Puff: Subjects inhaled P3L 50 µg/puff at the rate of one inhalation every 30 seconds on average, over approximately 6 minutes (i.e., 12 inhalations in total).
Arm/Group | P3L 50 µg/Puff
Number analyzed (Participants) | 15
ng/mL | 9.659 [6.724 to 13.874]

3. Primary Outcome: Maximum Concentration (Cmax) of Nicotine Following Single Use of P3L 80 µg/Puff
Description: T0 = start of product use.
  Derived from multiple blood sampling pre- and post-product use on Visit 5 (over 240 minutes post-product use).
  Geometric Least Squares (geometric LS) means are provided.
Time Frame: Visit 5: blood taken at 45, 30 and 15 minutes prior to T0 and 2, 4, 7, 10, 15, 20, 30, 40, 50, 60, 120, and 240 minutes after T0.
Population: PK population: all the subjects who have signed the informed consent, completed at least one P3L product use period and for whom at least one PK parameter can been derived.
  => 16 subjects - 1 subject withdrew after the product test at the admission visit - 1 subject discontinued by the Principal Investigator = 14 subjects
Measure: Least Squares Mean (95% Confidence Interval); unit: ng/mL
Groups:
- P3L 80 µg/Puff: Subjects inhaled P3L 80 µg/puff at the rate of one inhalation every 30 seconds on average, over approximately 6 minutes (i.e., 12 inhalations in total).
Arm/Group | P3L 80 µg/Puff
Number analyzed (Participants) | 14
ng/mL | 11.145 [7.701 to 16.128]

4. Primary Outcome: Maximum Concentration (Cmax) of Nicotine Following Single Use of P3L 150 µg/Puff
Description: T0 = start of product use.
  Derived from multiple blood sampling pre- and post-product use on Visit 6 (over 240 minutes post-product use).
  Geometric Least Squares (geometric LS) means are provided.
Time Frame: Visit 6: blood taken at 45, 30 and 15 minutes prior to T0 and 2, 4, 7, 10, 15, 20, 30, 40, 50, 60, 120, and 240 minutes after T0.
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: ng/mL
Groups:
- P3L 150 µg/Puff: Subjects inhaled P3L 150 µg/puff at the rate of one inhalation every 30 seconds on average, over approximately 6 minutes (i.e., 12 inhalations in total).
Arm/Group | P3L 150 µg/Puff
Number analyzed (Participants) | 14
ng/mL | 9.805 [6.775 to 14.189]

5. Primary Outcome: Time to the Maximum Concentration (Tmax) of Nicotine Following Single Use of Nicorette® Inhalator
Description: T0 = start of product use.
  Derived from multiple blood sampling pre- and post-product use on Visit 3 (over 240 minutes post-product use).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Nicorette® Inhalator
Number analyzed (Participants) | 15
minutes | 30.0 [20.0 to 40.0]

6. Primary Outcome: Time to the Maximum Concentration (Tmax) of Nicotine Following Single Use of P3L 50 µg/Puff
Description: T0 = start of product use.
  Derived from multiple blood sampling pre- and post-product use on Visit 4 (over 240 minutes post-product use).
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | P3L 50 µg/Puff
Number analyzed (Participants) | 15
minutes | 7.0 [4.0 to 7.0]

7. Primary Outcome: Time to the Maximum Concentration (Tmax) of Nicotine Following Single Use of P3L 80 µg/Puff
Description: T0 = start of product use.
  Derived from multiple blood sampling pre- and post-product use on Visit 5 (over 240 minutes post-product use).
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | P3L 80 µg/Puff
Number analyzed (Participants) | 14
minutes | 7.0 [7.0 to 7.0]

8. Primary Outcome: Time to the Maximum Concentration (Tmax) of Nicotine Following Single Use of P3L 150 µg/Puff
Description: T0 = start of product use.
  Derived from multiple blood sampling pre- and post-product use on Visit 6 (over 240 minutes post-product use).
Time Frame: as for outcome 4
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | P3L 150 µg/Puff
Number analyzed (Participants) | 14
minutes | 7.0 [4.0 to 7.0]

9. Primary Outcome: Area Under the Concentration-time Curve From Start of Product Use to the Last Quantifiable Time Point (AUC0-last) of Nicotine Following Single Use of Nicorette® Inhalator
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: h*ng/mL
Arm/Group | Nicorette® Inhalator
Number analyzed (Participants) | 15
h*ng/mL | 12.323 [9.251 to 16.415]

10. Primary Outcome: Area Under the Concentration-time Curve From Start of Product Use to the Last Quantifiable Time Point (AUC0-last) of Nicotine Following Single Use of P3L 50 µg/Puff
Description: as for outcome 2
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: h*ng/mL
Arm/Group | P3L 50 µg/Puff
Number analyzed (Participants) | 15
h*ng/mL | 9.943 [7.465 to 13.245]

11. Primary Outcome: Area Under the Concentration-time Curve From Start of Product Use to the Last Quantifiable Time Point (AUC0-last) of Nicotine Following Single Use of P3L 80 µg/Puff
Description: as for outcome 3
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: h*ng/mL
Arm/Group | P3L 80 µg/Puff
Number analyzed (Participants) | 14
h*ng/mL | 10.259 [7.644 to 13.770]

12. Primary Outcome: Area Under the Concentration-time Curve From Start of Product Use to the Last Quantifiable Time Point (AUC0-last) of Nicotine Following Single Use of P3L 150 µg/Puff
Description: as for outcome 4
Time Frame: as for outcome 4
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: h*ng/mL
Arm/Group | P3L 150 µg/Puff
Number analyzed (Participants) | 14
h*ng/mL | 9.983 [7.438 to 13.399]

13. Primary Outcome: Area Under the Concentration-time Curve From Start of Product Use to 10 Minutes After Start of Product Use (AUC0-10) of Nicotine Following Single Use of Nicorette® Inhalator
Description: as for outcome 1
Time Frame: Visit 3: blood taken at 45, 30 and 15 minutes prior to T0 and 2, 4, 7, and 10 minutes after T0.
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: h*ng/mL
Arm/Group | Nicorette® Inhalator
Number analyzed (Participants) | 15
h*ng/mL | 0.124 [0.077 to 0.200]

14. Primary Outcome: Area Under the Concentration-time Curve From Start of Product Use to 10 Minutes After Start of Product Use (AUC0-10) of Nicotine Following Single Use of P3L 50 µg/Puff
Description: as for outcome 2
Time Frame: Visit 4: blood taken at 45, 30 and 15 minutes prior to T0 and 2, 4, 7, and 10 minutes after T0.
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: h*ng/mL
Arm/Group | P3L 50 µg/Puff
Number analyzed (Participants) | 15
h*ng/mL | 1.028 [0.640 to 1.650]

15. Primary Outcome: Area Under the Concentration-time Curve From Start of Product Use to 10 Minutes After Start of Product Use (AUC0-10) of Nicotine Following Single Use of P3L 80 µg/Puff
Description: as for outcome 3
Time Frame: Visit 5: blood taken at 45, 30 and 15 minutes prior to T0 and 2, 4, 7, and 10 minutes after T0.
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: h*ng/mL
Arm/Group | P3L 80 µg/Puff
Number analyzed (Participants) | 14
h*ng/mL | 1.157 [0.714 to 1.874]

16. Primary Outcome: Area Under the Concentration-time Curve From Start of Product Use to 10 Minutes After Start of Product Use (AUC0-10) of Nicotine Following Single Use of P3L 150 µg/Puff
Description: as for outcome 4
Time Frame: Visit 6: blood taken at 45, 30 and 15 minutes prior to T0 and 2, 4, 7, and 10 minutes after T0.
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: h*ng/mL
Arm/Group | P3L 150 µg/Puff
Number analyzed (Participants) | 14
h*ng/mL | 1.040 [0.642 to 1.684]

ADVERSE EVENTS:
Time Frame: From the informed consent form (ICF) signature until the end of the safety follow-up period, up to 49 days (see the section "Detailed Description" for information on the study duration). The adverse events were tabulated for the safety population for: * Enrolment period (product test period, from enrolment to admission) * Nicorette® inhalator period * P3L 50 μg/puff period * P3L 80 μg/puff period * P3L 150 μg/puff period * Safety follow-up period
Description: The safety was assessed in the safety population, consisting of all subjects who have signed the ICF, and who have been exposed to P3L and/or Nicorette® inhalator.
  Safety population = 16 subjects.
  It should be noted that the assessment of clinical chemistry parameters occurred only at admission and Visit 6/early termination. Consequently, all safety laboratories occurring with product use where reported as pertaining to the last exposure period, i.e. P3L 150 μg/puff period.
Groups:
- Enrolment Period: All subjects who have signed the ICF, and who have been exposed to P3L and/or Nicorette® inhalator.
  Product test period - from enrolment to admission.
- Nicorette® Inhalator Period: Subjects inhaled the Nicorette® inhalator (15 mg) at the rate of one deep inhalation every 15 seconds on average, over approximately 20 minutes (80 inhalations in total).
- P3L 50 µg/Puff Period: Subjects inhaled P3L 50 µg/puff at the rate of one inhalation every 30 seconds on average, over approximately 6 minutes (i.e., 12 inhalations in total).
- P3L 80 µg/Puff Period: Subjects inhaled P3L 80 µg/puff at the rate of one inhalation every 30 seconds on average, over approximately 6 minutes (i.e., 12 inhalations in total).
- P3L 150 µg/Puff Period: Subjects inhaled P3L 150 µg/puff at the rate of one inhalation every 30 seconds on average, over approximately 6 minutes (i.e., 12 inhalations in total).
- Safety Follow-up Period: All subjects who have signed the ICF, and who have been exposed to P3L and/or Nicorette® inhalator entered a 7-day safety follow-up period during which (serious) adverse events can be spontaneously reported by the subjects.
Arm/Group | Enrolment Period | Nicorette® Inhalator Period | P3L 50 µg/Puff Period | P3L 80 µg/Puff Period | P3L 150 µg/Puff Period | Safety Follow-up Period
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15 | 0/15 | 0/14 | 0/14 | 0/16
Other Adverse Events (participants affected / at risk) | 7/16 | 3/15 | 4/15 | 4/14 | 8/14 | 2/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrolment Period (N=16) | Nicorette® Inhalator Period (N=15) | P3L 50 µg/Puff Period (N=15) | P3L 80 µg/Puff Period (N=14) | P3L 150 µg/Puff Period (N=14) | Safety Follow-up Period (N=16)
Blood Albumin Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Blood Triglycerides Increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood Glucose Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Blood Glucose Increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood Bilirubin Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood Cholesterol Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood Creatinine Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood Sodium Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 3 (3) | 3 (3) | 4 (4) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Skin Disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin Irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hot Flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
We confirm we have the contractual provisions in place which specify that in no event will the study site be allowed to disclose to any third party (or publicly release) any information obtained through the study without the CRO's prior written consent which in turn cannot provide such consent without Sponsor's approval unless such publication is made to satisfy regulatory requirements.

The Intellectual Property rights and research results from the present study belong to the Sponsor.